CLINICAL TRIAL: NCT00686335
Title: A New Modified-release Tablet Formulation of Prednisone (Lodotra®) in Patients With Nocturnal Asthma
Acronym: MONA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP01-201; EudraCT-Number: 2007-007316-29
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Results first posted 2012-12-28 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: asthma; nocturnal asthma; glucocorticoid dependent persistent asthma; signs and symptoms; lung function; prednisone
MeSH Terms: conditions — Asthma; Signs and Symptoms | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lodotra (Experimental): After the 4 week run-in period with immediate release prednisone (Cortancyl), patients were switched to the identical dose of modified release prednisone tablets (Lodotra). Study medication for the Lodotra treatment period consisted of Lodotra in 2 dose strengths (5 mg and 1 mg prednisone per tablet). Patients were to take their tablets with or after the evening meal (at 10 pm +/- 30 minutes) for 4 weeks.
  Interventions: Drug: Lodotra
- Cortancyl (Active Comparator): During the 4 week run-in period, patients remained on their respective pre-study dose of prednisone or equivalent. However, patients were standardized to 5 mg and 1 mg tablets of immediate release prednisone (Cortancyl). Patients were to take their tablets with or after the morning meal (at 8am +/- 30 minutes) for 4 weeks.
  Interventions: Drug: Cortancyl

INTERVENTIONS:
Drug: Lodotra — Administered with food at approximately 10 pm during the 4 week treatment period; patients received the identical dose of Lodotra as received of IR prednisone during the run-in period.
  Other Names: modified release tablet formulation of prednisone
  Arms: Lodotra
Drug: Cortancyl — Administered in the morning with food during the 4 week run-in period; patients remained on their respective pre-study dose of prednisone or equivalent standardized to 5 mg and 1 mg tablets of immediate release (IR) prednisone (Cortancyl).
  Other Names: immediate release prednisone tablets
  Arms: Cortancyl

SUMMARY:
The purpose of the study is to evaluate in subjects suffering from nocturnal asthma, the efficacy and safety of modified release Prednisone on signs and symptoms.

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be able to understand the terms of the written informed consent form, and must provide a dated and signed form before the start of any study procedure
* At least 18 years old
* Patient having a diagnosis of asthma dating back more than 6 months at the time of inclusion
* Asthma necessitating a continuous treatment by oral corticoids
* A minimum of 3 nocturnal awakenings due to asthma during the last screening week
* Stable dose of oral glucocorticoids for at least 4 weeks prior to inclusion into the study
* No change in asthma medication during the last 4 weeks prior to V0
* Non-smoker or ex-smoker (having stopped smoking more than one year previously and with a smoking history of less than 10 pack years )
* Female patients of childbearing potential must be using a medically accepted contraceptive regimen
* Able to perform the required study procedures including handling of medication containers and diaries

Exclusion Criteria:

* Poorly controlled asthma, defined as meeting at least one of the following within the 4 weeks prior to Visit V0:

  * hospital admission for asthma (including treatment in an emergency room),
  * a lower airway infection,
* Diagnosis of chronic obstructive pulmonary disease or other relevant lung diseases (e.g. history of bronchiectasis, cystic fibrosis, bronchiolitis, lung resection, lung cancer, active tuberculosis, interstitial lung disease)
* Clinically significant abnormalities of the hematological or biochemical constants
* Pregnancy or breastfeeding
* Participation in another clinical study within 30 days preceding Visit V0,
* Re-entry of patients previously enrolled in this trial,
* Suspected inability or unwillingness to comply with the study procedures
* Alcohol or drug abuse
* Need to take a non-authorised concomitant treatment (cf. list of medicaments not authorised during the study) in the course of the study
* Other disease requiring treatment with corticosteroids
* Subject is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Patient with a hospitalisation scheduled during the study period
* Any uncontrolled concomitant disease requiring further clinical evaluation (e.g. uncontrolled diabetes, uncontrolled hypertension, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel MD, Study Director — Amgen
Locations (1):
- Hôpital Bichat, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Asthmatic patients, aged at least 18 years, suffering from severe persistent asthma, having nocturnal symptoms and receiving treatment with oral glucocorticoids were recruited from Hôpital Bichat between July 2008 and March 2010.
Pre-assignment Details: After a 4-week run-in period in which patients were treated with immediate release prednisone (Cortancyl®) administered in the morning, all eligible patients (based on inclusion/exclusion criteria) were treated for 4 weeks with an identical dose of Lodotra administered in the evening.
Groups:
- Safety Population: all patients that started the run-in period with Cortancyl®
Period: Run-in Period
Arm/Group | Safety Population
Started | 12
Completed | 7
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — asthma exacerbation | 1
Not completed — violation of inclusion/exclusion criteri | 3
Period: Treatment Period
Arm/Group | Safety Population
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Safety Population
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (14.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  France | 12

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Nocturnal Awakenings During the Last 2 Weeks of Treatment
Description: Variation in the total number of nocturnal awakenings during the last 2 weeks of run-in treatment with Cortancyl and the last 2 weeks of treatment with Lodotra.
Time Frame: 4 weeks and 8 weeks
Population: The efficacy analysis population included all 7 patients who completed both study periods without major protocol deviations.
Measure: Mean (Standard Deviation); unit: number of nocturnal awakenings
Groups:
- Lodotra: modified release prednisone
- Cortancyl: immediate release prednisone
Arm/Group | Lodotra | Cortancyl
Number analyzed (Participants) | 7 | 7
number of nocturnal awakenings | 2.1 (4.41) | 10.0 (5.45)
Statistical Analysis 1: Comparison: Lodotra vs Cortancyl; As this was an explorative study to collect data for a subsequent controlled study, no hypothesis testing was performed. All analyses were descriptive; Test type: Superiority or Other; Other — As this was an explorative study to collect data for a subsequent controlled study, no hypothesis testing was performed. All analyses were descriptive; As this was an explorative study, no hypothesis testing was performed. All analyses were descriptive; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-13.5 to -2.2], Standard Deviation 6.07

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the patient gave informed consent until the end of the follow-up visit or 30 days after last study drug administration, whichever occurred later.
Description: Safety was evaluated by:
  * recording of Adverse Events (AEs) and concomitant treatments at each visit
  * physical examination and vital sign measurements at each visit
  * laboratory safety assessments at visits V0 and V4
Arm/Group | Lodotra | Cortancyl
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/12
Other Adverse Events (participants affected / at risk) | 6/7 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lodotra (N=7) | Cortancyl (N=12)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — 1 patient experienced 2 Serious Adverse Events (SAEs). Respiratory deterioration developed during run-in period;pt was withdrawn from study. 4 days later, pt experienced an asthma exacerbation and was hospitalized. The patient recovered.
arterial thrombosis (Vascular disorders) | 0 | 1 — One patient experienced 2 serious adverse events. Arteritis was a baseline event which became serious during the run-in period due to hospitalization. Patient was discontinued from the study, surgery was performed, and patient recovered.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lodotra (N=7) | Cortancyl (N=12)
asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
insomnia (Psychiatric disorders) | 2 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hernial eventration (Gastrointestinal disorders) | 1 | 0
influenza like illness (General disorders) | 1 | 1
menstrual disorder (Reproductive system and breast disorders) | 1 | 0
oedema (General disorders) | 1 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
tremor (Nervous system disorders) | 1 | 0
tooth extraction (Surgical and medical procedures) | 1 | 0
anxiety (Psychiatric disorders) | 0 | 1
bronchitis (Infections and infestations) | 0 | 3
fungal skin infection (Infections and infestations) | 0 | 1
haematoma (Vascular disorders) | 0 | 1
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
sinusitis (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
This was an explorative study to collect data for a subsequent controlled trial and therefore no hypothesis testing was performed. The size of the efficacy population (N=7) is too small to detect any statistically significant changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Anything concerning publication, information and communication is described under law number R5121-13 of the French Code de la Santé Publique. Any information about results cannot be given without the accordance of Horizon Pharma (formerly Nitec Pharma).